CLINICAL TRIAL: NCT03128801
Title: Effects of Self-Stretching Posture and Segmental Stabilization on Pain and Disability in Patients With Chronic Low Back Pain: Randomized Controlled Trial and Blinded
Brief Title: Effects of Self-Stretching Posture and Segmental Stabilization in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thais Cristina Chaves, Professor, Department of Neuroscience and Behavioral Science at the Ribeirão Preto Medical School at the University of Sao Paulo. Coordinator, Laboratory of Interdisciplinary Research on Musculoskeletal Pain., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 045641
Record Dates: First submitted 2017-04-10; First posted 2017-04-25 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Back Pain; Muscle Stretching Exercises; Stabilization Exercise; Exercise Therapy; Exercise Movement; Exercise Movement Tecniques; Pain; Disability
MeSH Terms: conditions — Low Back Pain; Back Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global Stretching Program (GSP) (Experimental): Participants will be submitted to a GSP in self-management postures weekly for 40 minutes session conducted by one one physical therapist, certified to use the technique (Stretching Global Active).
  Interventions: Procedure: Global Stretching Program
- Stabilization Exercises (Active Comparator): A exercise protocol will be administered and the criteria to increase exercise progression was previously described by Hicks et al (2005).
  Interventions: Procedure: Stabilization Exercises

INTERVENTIONS:
Procedure: Global Stretching Program — Participants will be submitted to a GSP in self-management postures weekly for 40 minutes session conducted by one one physical therapist, certified to use the technique (Stretching Global Active). The GSP will last for a period of 8 weeks. The protocol is based on the study of Lawand et al (2015) who used all postures global therapeutic stretching. The investigators will use six self-management postures in a standardized manner, each of which will last for 10 to 20 minutes.
  Arms: Global Stretching Program (GSP)
Procedure: Stabilization Exercises — The exercise protocol and criteria to increase exercise progression was previously described by Hicks et al (2005). It will be directed by a single therapist one to one session based on specific criteria (being able to maintain muscle contraction eight seconds during 30 repetitions in bilateral exercises or during 20 repetitions for unilateral exercises). Each session will be conducted weekly for 40 minutes.
  Arms: Stabilization Exercises

SUMMARY:
Background: Low back pain is a major problem for public health that affects about 60-85% of the population at some point in life. Approximately 10-40% of individuals with low back pain develop the chronic form. International guidelines consider three groups of treatment options for low back pain: medication, invasive and conservative treatments in which conservative approach is the most recommended. The European Guidelines for Management of Chronic Non-specific Low Back Pain recommends that supervised exercise programs should be used as front-line treatment for chronic low back pain, such as stabilization exercises, conventional stretching and other active exercise, but there is no consensus on literature on the most effective form of treatment. However, there is limited evidence about the effects of a global stretching intervention using self-stretching postures for chronic low back pain.

Objectives: The aim of this research is to compare the effects of an active global stretching program (GSP) using self-management of posture versus stabilization exercises on pain intensity and disability for patients with chronic non-specific low back pain.

Methods: This study is a randomized controlled three arm clinical trial with examiner blinding. A sample of 100 patients with chronic non-specific low back pain will be randomly assigned to two treatment groups (GSP or Stabilization Exercises). The eligibility criteria will be 18 and 50 years, pain in the last three months and/or pain in at least half of the days in the past six months, pain located between T12 and the gluteal folds, pain intensity greater than or equal to three, and score greater than 14% on Oswestry Disability Index. Patients will be assessed in baseline, immediately after treatment and after one and three-months follow-up. Sessions will be provided weekly for eight weeks by a single therapist lasting 40 minutes. The primary outcomes will be pain intensity and low back pain related disability and the secondary outcomes will be fear avoidance, global perceived effect of treatment and muscle flexibility. All statistical analysis will be conducted following principles of intention to treat, and the treatment effects will be calculated using linear mixed models.

DETAILED DESCRIPTION:
Study design

This study will be a randomized controlled with two arm clinical trial and examiner blinding.

The sample will consist of 100 participants (both genders) with nonspecific chronic low back pain.

Randomization and allocation

Patients will be randomly assigned through a randomization process involving opaque envelopes containing cards stipulating one of the three following groups: (1) Global Stretching Program (GSP) and (2) Stabilization Exercises (SE). An assistant researcher not involved in the recruitment of patients will allocate the randomly using data generated by a group allocation software.

Procedures

The proposed study will follow the recommendations described on Consolidated Standards of Reporting Trials (CONSORT) statement to ensure transparency and quality of the findings.

Each participant will be supervised by a single physical therapist, who will not be involved in the assessment of the patients and/or randomization. A second researcher will conduct the following evaluation in baseline assessment: pain intensity, low back pain related disability and psychosocial factors using questionnaires validated to Brazilian Portuguese.

During the treatment and follow-up periods, the use of drugs will be discouraged. Patients who require rescue medication during the study will be encouraged to register the use.

Initial evaluation and follow-up

After eligibility assessment, participants will be asked to complete a questionnaire with personal data. Subsequently, the psychosocial evaluation will be conducted in accordance with the recommendations of the Initiative on Methods, Measurement and Pain Assessment in Clinical Trials (IMMPACT) for chronic pain. The volunteers will be re-assessed immediately after treatment and after one and three-months follow-up. The main outcome measures will be pain intensity and low back pain related disability. Secondary outcomes will be fear avoidance, global perceived treatment effect and muscle flexibility.

The hypothesis of this study is that patients with chronic low back pain submitted to global stretching exercises will show greater effects to pain intensity and disability than patients submitted to interventions separated.

Primary Outcomes

The pain intensity measurement will be accomplished by application of a numerical pain rating scale - PNRS, which consists of a sequence of eleven numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable". Volunteers will rate their pain based on these parameters.

To assess disability related to chronic low back pain, the Oswestry Low Back Disability Index, adapted to Brazilian Portuguese will be used. The result is converted into a percentage by multiplying the total score by two. This instrument consists of 10 items, each of which has six response options. The total score will be calculated by summing up the points, the largest possible sum being #50. Previous research has found ODI showed responsiveness to change for patients with CLBP, with MCID of #8 points.

Secondary Outcomes

Fingertip-to-Floor Test, Fear avoidance beliefs questionnaire - FABQ and Global Perceived Effect of Treatment will be assessed pre and post treatment.

The FABQ adapted for Brazilian Portuguese consists of 16 self- response items, rated on a seven-point Likert scale from 0 (completely disagree) to 6 (completely agree). The score is obtained for each separate subscale: one that addressed the fears and beliefs of individuals in relation to work and one that addressed their fears and beliefs about physical activities.

Global Perceived Effect of Treatment is recommended for use in clinical trials of chronic pain as a measure of the perception of global improvement/worsening regarding to treatment. Global Perceived Effect of Treatment is an 11-point scale that ranges from -5 ("vastly worse") through 0 ("no change") to +5 ("completely recovered"). A higher score indicates higher recovery from the condition.

The Fingertip-to-floor test showed excellent levels of validity compared to the radiological measurement (r=0.96) and reproducibility (intra and interexaminer - ICC = 0.99). The test is known for full mobility in the tilted forward position when standing, corresponding to flexion of the spine and pelvis. It is a measure of relevance in rehabilitation results probably because patients simultaneously increase the pelvic and lumbar flexion post treatment.

As baseline intervention the investigators will assess pain catastrophising, anxiety and depression scale and pain self efficacy. Hospital Anxiety and Depression Scale will be used to identify anxiety disorders and depression in physically ill patients. The HADS was translated and validated into Portuguese. Then divided into the anxiety subscale (HADS-A) and the depression subscale (HADS-D), both containing seven interspersed items. It is composed of seven items for depression and seven items for anxiety, each item including four response options ranging from 0 to 3. The cutoff scores are 8 points for anxiety, 9 for depression. Change in depressive symptoms significantly predicted change in pain severity and intensity.

Pain catastrophising scale (PCS) will be used to assess catastrophising thoughts. The scale is composed of 13 items staggered on a Likert scale, ranging from 0 to 5 points. The total score is the sum of the items divided by the number of items answered, with the minimum score being 0 and the maximum being 5 for each item. Higher scores indicated a greater presence of catastrophic thoughts. The total score of the scale could vary between 0 and 52 points. A recent systematic review found that found catastrophising to be associated with pain and disability at follow-up in CLBP patients.

The Chronic Pain Self-Efficacy Scale (CPSS) will be used to assess self-efficacy perception related to chronic pain, which can be defined as an individual's personal conviction that they can successfully execute an action to produce desirable results related to living with chronic pain. The scale has 22 items and was adapted and validated to Brazilian Portuguese. Previous research suggested that rehabilitation programs for CLBP should target pain self-efficacy which mediates the relationship between depressive symptoms and pain severity.

Interventions

Participants will be randomly assigned to two possible interventions: GPS and Stabilization Exercises intervention group. Treatment protocol will be conducted by eight weeks, one time per week. The session will last for 40 minutes.

Data Analysis

The pain intensity outcome was considered for sample size calculation. A change of at least 2 units on NPRS was considered for analysis. The sample size obtained was 78 (39 subjects each). The following specifications were considered: α = 5%, statistical power of 90% and 0.61 effect size for F-test. The GPower software was used to calculate the sample size (GPower 3.0.10 of the University of Kiel, Germany). Thus, to ensure a power suitable and assuming sample losses, 100 (50 subjects per group) participants will be considered (GPower 3.0.10, University of Kiel, Germany).

The statistician will be given grouped data, but data will be coded so that the statistician will remain blinded to patients' group allocation and to protect patient confidentiality. The mean effects of the interventions and the group differences for all outcomes (primary and secondary) will be calculated using linear mixed models that incorporated terms for the treatment groups, time (post-intervention and follow-up), and interaction terms (treatment subgroups and time) as well as psychosocial variables, sex and age as covariates. Secondary analysis will be conducted using regression models to determine whether baseline scores of psychosocial variables (HADS, PCS, CPSS) will moderate the effect of treatments. The analyzes will follow the intention-to-treat principles. For all of these analyzes, IBM SPSS software package will be used, version 22 (IBM Corp, New York).

The Statistical Package for the Social Sciences (SPSS) software version 22 (Chicago, IL, USA) will be used for analysis, and the significance level was established at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 60 years;
* medical diagnosis of chronic non-specific low back pain in the last 3 months and/or pain during at least half of the days in the past 6 months (Deyo et al. 2014), that is located between T12 and the gluteal folds;
* pain intensity equal to or greater than three;
* pain caused by certain postures, activities and movements; and
* score greater than 14% on the Oswestry Lumbar Disability Index (Vibe Fersum et al. 2013)

Exclusion Criteria:

* red flags (neoplastic diseases or tumors in the spine, inflammatory diseases, infections and fractures);
* serious neurological (or central and peripheral neurological) symptoms, psychiatric, rheumatologic and cardiac diseases;
* acute radiculopathy;
* lumbar stenosis;
* spondylolisthesis;
* history of spinal surgeries;
* pregnancy; and
* underwent physical therapy treatments (less than 6 months before the evaluation period).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Immediately after
  The pain intensity measurement will be accomplished by application of a numerical pain rating scale - NPRS which consists of a sequence of eleven numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable". Volunteers will rate their pain based on these parameters.
Low Back Pain related-Disability | Immediately after
  To assess disability related to chronic low back pain, the Oswestry Low Back Disability Index - ODI, adapted to Brazilian Portuguese will be used. The result is converted into a percentage by multiplying the total score by two. This instrument consists of 10 items, each of which has six response options. The total score will be calculated by summing up the points, the largest possible sum being #50. Previous research has found ODI showed responsiveness to change for patients with CLBP.

SECONDARY OUTCOMES:
Fear avoidance beliefs questionnaire (FABQ) | Immediately after
  The FABQ adapted for Brazilian Portuguese, consists of 16 self- response items, rated on a seven-point Likert scale from 0 (completely disagree) to 6 (completely agree). The score is obtained for each separate subscale: one that addressed the fears and beliefs of individuals in relation to work and one that addressed their fears and beliefs about physical activities.
Global Perceived Effect of Treatment | Immediately after
  Global Perceived Effect of Treatment is recommended for use in clinical trials of chronic pain as a measure of the perception of global improvement/worsening regarding to treatment. Global Perceived Effect of Treatment is an 11-point scale that ranges from -5 ("vastly worse") through 0 ("no change") to +5 ("completely recovered"). A higher score indicates higher recovery from the condition.
Fingertip-to-Floor Test | Immediately after
  The Fingertip-to-floor test showed excellent levels of validity compared to the radiological measurement (r=0.96) and reproducibility (intra and interexaminer - ICC = 0.99). The test is known for full mobility in the tilted forward position when standing, corresponding to flexion of the spine and pelvis. It is a measure of relevance in rehabilitation results probably because patients simultaneously increase the pelvic and lumbar flexion post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Thais C Chaves, Professor, Study Chair — University of São Paulo - Ribeirao Preto School of Medicine
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The results will be available in manuscripts published in peer reviewed journals.

REFERENCES:
- [Derived] Turci AM, Nogueira CG, Nogueira Carrer HC, Chaves TC. Self-administered stretching exercises are as effective as motor control exercises for people with chronic non-specific low back pain: a randomised trial. J Physiother. 2023 Apr;69(2):93-99. doi: 10.1016/j.jphys.2023.02.016. Epub 2023 Mar 21. PMID 36958977